CLINICAL TRIAL: NCT04079933
Title: A Randomized, Controlled, Parallel Group Clinical Study of Cigarette Smokers Using an Innovative Oral Tobacco-derived Nicotine Product to Determine Impact on Cigarette Consumption and Biomarkers of Exposure
Brief Title: A Study to Evaluate Changes in Smokers Using An Oral Tobacco-Derived Nicotine Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altria Client Services LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COV-VER-01-13
Record Dates: First submitted 2019-08-14; First posted 2019-09-06 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-05

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Continue Smoking (No Intervention): Subjects were asked to continue smoking their own brand of cigarettes ad libitum for 4 weeks
- Group 2: OTDN (Experimental): Subjects were allowed to continue smoking their own brand of cigarettes ad libitum and provided the option to use an OTDN (specifically, VERVE® Discs Blue Mint [VBM-FG2]) also under ad libitum conditions
  Interventions: Other: Oral tobacco-derived nicotine product (OTDN)

INTERVENTIONS:
Other: Oral tobacco-derived nicotine product (OTDN)
  Other Names: VERVE® Discs Blue Mint, VBM-FG2 oral discs
  Arms: Group 2: OTDN

SUMMARY:
The purpose of this study was to estimate changes in biomarkers of exposure (BOE) in adult cigarette smokers using an oral tobacco-derived nicotine (OTDN) product relative to adult smokers who continue smoking exclusively.

DETAILED DESCRIPTION:
This was a randomized, controlled, open-label, parallel group, multicenter, 9-week study to determine changes in BOE in adult smokers allowed ad libitum use of an OTDN product relative to adult smokers who were not allowed to use an OTDN product. This study was conducted in adult smokers who were considered to be in overall good health. Subjects were randomized to Test (allowed OTDN use) or Control (not allowed OTDN use) groups.

ELIGIBILITY:
Inclusion Criteria:

Subject must:

1. sign an Institutional Review Board (IRB)-approved Informed Consent Form (ICF) for the study.
2. be between the ages of 21 and 65 years, inclusive, at the time of Screening.
3. have consumed a minimum of 10 manufactured cigarettes per day (CPD) daily during the last 6 months (entire 6 month period must have occurred after subject turned 21 years of age).
4. indicate that he/she smokes cigarettes "every day" at Screening and on Day 1
5. be able to fully comprehend the English language.
6. have an active phone number and must have daily access to a touchtone phone between 1600 and 1900 hours.
7. be interested in alternative tobacco products to cigarettes at Screening.
8. indicate that they "definitely would buy" or "probably would buy" on the VBM-FG2 Potential Purchase Interest Questionnaire.
9. be in generally good health.
10. if female, have a negative urine dipstick pregnancy test.
11. if female heterosexually active and of childbearing potential (i.e., not surgically sterile or two years naturally postmenopausal), agree to use a medically accepted method of contraception from Screening through the End of Study.
12. have clinical laboratory tests within the appropriate reference range or which are clinically acceptable to the Investigator.
13. have a negative ethanol, amphetamines, opiates, cannabinoids, and cocaine urine drug screen.
14. test negative for human immunodeficiency (HIV), hepatitis B (hepatitis B surface antigen [HBsAg]), and Hepatitis C (anti-hepatitis C virus antibody [anti-HCV]).
15. be willing and able to comply with the requirements of the study.

Exclusion Criteria:

Subject must not:

1. be pregnant, nursing, or planning to become pregnant during the study period.
2. indicate that he/she intends to quit smoking within the next 30 days (at Screening or on Day 1).
3. have uncontrolled hypertension, history of coronary heart disease or other significant heart conditions, and/or other significant medical conditions that might interfere with study procedures.
4. have used prescription anti-diabetic medication and/or insulin therapy within 12 months of Day 1.
5. have a history of drug or alcohol abuse within the 24 months prior to Screening.
6. have participated in a clinical study for an investigational drug, device, or biologic within 30 days prior to enrollment (Day 1).
7. be a current user of nicotine replacement therapy (indicate every day or some days on Subject Screener/Tobacco History Questionnaire).
8. be a current or former employee of the tobacco industry or a first-degree relative (e.g., parent, sibling, child) of a current or former employee of the tobacco industry.
9. have been involved in the development of the study design/conduct or be a first-degree relative (e.g., parent, sibling, child) of someone involved in the development of the study design/conduct.
10. be a current employee or personnel involved with the study at the study site.
11. be currently participating in the study at a different study site (i.e., each subject can only be in the study population once).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study enrolled adult male and female (no more than 60% of either gender) self-affirmed combustible cigarette smokers
Enrollment: 154 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2013-11-26 (Actual); Study Completion 2013-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery S Edmiston, PhD, Study Director — Altria Client Services LLC
Locations (3):
- United States (3):
  - Covance Daytona Clinical Research Unit, Daytona Beach, Florida
  - Covance Evansville Clinical Research Unit, Evansville, Indiana
  - Covance Dallas Clinical Research Unit, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were required to complete an 8 day baseline assessment during which subject cigarette use data was collected using daily interactive voice response system (IVRS) calls and recall of the previous week methods. Three subjects were withdrawn from the study prior to randomization. A total of 154 subjects were randomized in this study; 92 subjects were randomized to the Test Group and 62 subjects were randomized to the Control Group.
Groups:
- Test (ad Libitum VERVE® Discs Blue Mint [VBM-FG2] Use): Subjects were allowed to continue smoking their own brand of cigarettes ad libitum and were provided the option to use the test product (VBM-FG2 oral discs) also under ad libitum conditions.
- Control (no VBM-FG2): Subjects were asked to continue smoking their own brand of cigarettes ad libitum for 4 weeks
Period: Overall Study
Arm/Group | Test (ad Libitum VERVE® Discs Blue Mint [VBM-FG2] Use) | Control (no VBM-FG2)
Started | 92 | 62
Completed | 89 | 57
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Test (ad Libitum VBM-FG2): Subjects were allowed to continue smoking their own brand of cigarettes ad libitum and were provided the option to use the test product (VBM-FG2 oral discs) also under ad libitum conditions
- Total: Total of all reporting groups
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2) | Total
Number analyzed (Participants) | 92 | 62 | 154
Age, Continuous [Mean (Full Range); unit: years] | 43 [21 to 65] | 42 [21 to 64] | 43 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 30 | 78
  Male | 44 | 32 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 86 | 59 | 145
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 0 | 1
  Race: Black or African American | 15 | 11 | 26
  Race: White | 72 | 47 | 119
  Race: Other | 4 | 4 | 8
Body Weight [Mean (Standard Deviation); unit: kg] | 82.8 (20.94) | 85.3 (23.56) | 83.8 (21.99)
Height [Mean (Standard Deviation); unit: cm] | 170.8 (8.32) | 171.1 (9.40) | 170.9 (8.75)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.3 (6.69) | 29.0 (7.26) | 28.6 (6.91)
Quit Attempts [Count of Participants; unit: Participants] — Quit Attempts and Quitting Intentions Questionnaire - Day 1 was used to determine Quit Attempts
  Participants
    Yes | 3 | 3 | 6
    No | 89 | 59 | 148
Cigarette Consumption per Day [Count of Participants; unit: Participants] — Day 7 IVRS data (or the last available data entered before the Day 8 site visit) were used to derive the Cigarette Consumption per day and it was in the randomization on Day 8
  Participants
    ≤ 20 | 66 | 44 | 110
    >20 | 26 | 18 | 44
Quit Attempts in previous 6 months [Mean (Standard Deviation); unit: smoking cessations] — Number of times stopped smoking cigarettes for 24 hours or longer in an attempt to quit in past 6 months Population: Intent to Treat population. Data was not available for four subjects.
  smoking cessations
    number analyzed (Participants) | 89 | 61 | 150
    (all) | 0.3 (0.89) | 0.2 (0.67) | 0.3 (0.81)
Number of years smoked since turning 21 years of age [Mean (Standard Deviation); unit: years] — Population: Intent to Treat population. Data was not available for three subjects.
  years
    number analyzed (Participants) | 91 | 60 | 151
    (all) | 19.5 (10.99) | 20.3 (10.30) | 19.8 (10.69)

OUTCOME MEASURES:

1. Primary Outcome: Summary Statistics of Percent Change From Baseline for Urinary Total 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) (%) (Per-Protocol Population)
Description: Summary statistics of percent change from baseline for urinary total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol [NNAL] (%) in each study visit are presented.
  Baseline taken from Visit 3 (Day 8±1) value. Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
  Mean percent change from baseline is the mean of all individual subjects' percent change from baseline values. Each percent change from baseline was calculated by subtracting the individual subject's baseline value from the value at the desired timepoint and then dividing this calculated value by the individual subject's baseline value and multiplying by 100. These individual subjects' percent changes from baseline values were used to calculate the mean percent change from baseline using a Statistical Analysis System (SAS®) procedure.
Time Frame: Day 15 (Visit 4), Day 22 (Visit 5), Day 29 (Visit 6) and Day 36 (Visit 7/End of Study) relative to the start of the baseline period (Visit 2/Day 1)
Population: Per-protocol population. All Per-Protocol Test and Control subjects were included in the analysis. If a value was missing for any subject at any visit, that subject's value was omitted from the analysis for that visit only.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
percent change from baseline
  Visit 4: number analyzed (Participants) | 80 | 53
  Visit 4 | 3.8 (34.11) | 13.8 (45.56)
  Visit 5: number analyzed (Participants) | 83 | 51
  Visit 5 | 12.5 (60.16) | 30.4 (63.66)
  Visit 6: number analyzed (Participants) | 79 | 53
  Visit 6 | 16.0 (50.87) | 29.2 (46.70)
  End of Study/Early Termination: number analyzed (Participants) | 84 | 54
  End of Study/Early Termination | 15.4 (62.42) | 28.4 (57.66)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline in urinary total NNAL; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline in urinary total NNAL; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline in urinary total NNAL; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline in urinary total NNAL; p = 0.2347, t-test, 2 sided; Mean Difference (Net) = -12.6, 95% CI 2-sided [-33.5 to 8.27] — Difference in Least Square (LS) means (Test - Control) using Mixed Effects Repeated Measures Model 1: Percent Change from baseline = study group + visit + study group*visit + subject + random error, fitted with unstructured covariance matrix
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.2905, t-test, 2 sided; Mean Difference (Net) = -11.9, 95% CI 2-sided [-33.9 to 10.2] — Difference in LS means (Test - Control) using Mixed Effects Repeated Measures Model 2: %Change from baseline = study group +visit +study group*visit +CPD +Sex +Race +BMI +Age +subject +random error, fitted with unstructured covariance matrix

2. Secondary Outcome: Summary Statistics of Change From Baseline for Urinary Total NNAL (ng/g Creatinine) (Per-Protocol Population)
Description: Summary statistics of change from baseline for urinary total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol [NNAL] (ng/g creatinine) in each study visit are presented.
  Baseline taken from Visit 3 (Day 8±1) value. Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
ng/g
  Visit 4: number analyzed (Participants) | 80 | 53
  Visit 4 | 14.99 (212.505) | 9.47 (207.308)
  Visit 5: number analyzed (Participants) | 83 | 51
  Visit 5 | 70.90 (436.326) | 76.50 (310.423)
  Visit 6: number analyzed (Participants) | 79 | 53
  Visit 6 | 66.23 (303.806) | 117.69 (289.763)
  End of Study/Early Termination: number analyzed (Participants) | 84 | 54
  End of Study/Early Termination | 81.33 (345.110) | 86.53 (209.749)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in urinary total NNAL; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline to end of study in urinary total NNAL; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in urinary total NNAL; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline to end of study in urinary total NNAL; p = 0.9433, t-test, 2 sided; Mean Difference (Net) = -3.72, 95% CI 2-sided [-107 to 99.4] — Difference in LS means (Test - Control) using Mixed Effects Repeated Measures Model 1: Change from baseline = study group + visit + study group*visit + subject +random error, fitted with unstructured covariance matrix
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in urinary total NNAL; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in urinary total NNAL; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in urinary total NNAL; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in urinary total NNAL; p = 0.8264, t-test, 2 sided; Mean Difference (Net) = -12.2, 95% CI 2-sided [-122 to 97.5] — Difference in LS means (Test - Control) using Mixed Effects Repeated Measures Model 2: Change from baseline= study group + visit + study group*visit + CPD + Sex + Race + BMI + Age + subject + random error, fitted with unstructured covariance matrix

3. Secondary Outcome: Summary Statistics of Change From Baseline for Nicotine Equivalents (mg / g Creatinine) (Per-Protocol Population)
Description: Summary statistics of change from Baseline for urinary nicotine equivalents including nicotine and its 5 metabolites (cotinine, trans-3'-hydroxycotinine, trans-3'-hydroxycotinine-0-glucuronide, nicotine-N-glucuronide, and cotinine-N-glucuronide) (mg/g creatinine) in each study visit are presented.
  Baseline taken from Visit 3 (Day 8±1) value. Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
mg/g
  Visit 4: number analyzed (Participants) | 70 | 47
  Visit 4 | -0.6 (5.28) | 0.6 (6.45)
  Visit 5: number analyzed (Participants) | 74 | 43
  Visit 5 | 1.9 (8.46) | 2.5 (6.48)
  Visit 6: number analyzed (Participants) | 66 | 46
  Visit 6 | 1.1 (8.03) | 4.3 (9.47)
  End of Study/Early Termination: number analyzed (Participants) | 74 | 46
  End of Study/Early Termination | 2.6 (9.75) | 3.6 (6.89)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in nicotine equivalents; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in nicotine equivalents; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in nicotine equivalents; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in nicotine equivalents; p = 0.4903, t-test, 2 sided; Mean Difference (Net) = -1.13, 95% CI 2-sided [-4.35 to 2.10] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.4251, t-test, 2 sided; Mean Difference (Net) = -1.40, 95% CI 2-sided [-4.88 to 2.07] — [estimate comment as in outcome 2, analysis 2]

4. Secondary Outcome: Summary Statistics of Percent Change From Baseline for Nicotine Equivalents (%) (Per-Protocol Population)
Description: Summary statistics of percent change from Baseline for urinary nicotine equivalents including nicotine and its 5 metabolites (cotinine, trans-3'-hydroxycotinine, trans-3'-hydroxycotinine-0-glucuronide, nicotine-N-glucuronide, and cotinine-N-glucuronide) (%) in each study visit are presented.
  Baseline taken from Visit 3 (Day 8±1) value. Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
  Mean percent change from baseline is the mean of all individual subjects' percent change from baseline values. Each percent change from baseline was calculated by subtracting the individual subject's baseline value from the value at the desired timepoint and then dividing this calculated value by the individual subject's baseline value and multiplying by 100. These individual subjects' percent changes from baseline values were used to calculate the mean percent change from baseline using a SAS® procedure.
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
percent change from baseline
  Visit 4: number analyzed (Participants) | 70 | 47
  Visit 4 | 3.2 (37.85) | 14.8 (51.81)
  Visit 5: number analyzed (Participants) | 74 | 43
  Visit 5 | 18.7 (57.95) | 26.3 (50.78)
  Visit 6: number analyzed (Participants) | 66 | 46
  Visit 6 | 15.7 (54.02) | 30.8 (53.08)
  End of Study/Early Termination: number analyzed (Participants) | 74 | 46
  End of Study/Early Termination | 25.2 (65.08) | 35.5 (60.54)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study in nicotine equivalents; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study in nicotine equivalents; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study in nicotine equivalents; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study in nicotine equivalents; p = 0.4060, t-test, 2 sided; Mean Difference (Net) = -9.83, 95% CI 2-sided [-33.2 to 13.5] — Difference in Least Square means (Test - Control) using Mixed Effects Repeated Measures Model 1: Percent Change from baseline = study group + visit + study group*visit + subject + random error, fitted with unstructured covariance matrix
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 4, analysis 1]; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.4165, t-test, 2 sided; Mean Difference (Net) = -10.3, 95% CI 2-sided [-35.4 to 14.7] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Summary Statistics of Change From Baseline for S-phenyl Mercapturic Acid (S-PMA) (ng/g Creatinine) (Per-Protocol Population)
Description: Summary statistics of change from Baseline for urinary S-phenyl mercapturic acid [S-PMA] (ng/g creatinine) in each study visit are presented.
  Baseline taken from Visit 3 (Day 8±1) value. Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
ng/g
  Visit 4: number analyzed (Participants) | 79 | 50
  Visit 4 | 506.33 (3150.049) | 242.66 (2846.817)
  Visit 5: number analyzed (Participants) | 82 | 49
  Visit 5 | 1129.88 (4867.996) | 809.04 (3649.614)
  Visit 6: number analyzed (Participants) | 74 | 51
  Visit 6 | 1102.42 (4045.946) | 1637.29 (4348.050)
  End of Study/Early Termination: number analyzed (Participants) | 81 | 51
  End of Study/Early Termination | 903.49 (4985.072) | 1160.48 (2798.644)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in S-PMA; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in S-PMA; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in S-PMA; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in S-PMA; p = 0.7240, t-test, 2 sided; Mean Difference (Net) = -269, 95% CI 2-sided [-1773 to 1235] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 5, analysis 1]; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; p = 0.9508, t-test, 2 sided; Mean Difference (Net) = 50.5, 95% CI 2-sided [-1566 to 1667] — [estimate comment as in outcome 2, analysis 2]

6. Secondary Outcome: Summary Statistics of Percent Change From Baseline for S-PMA (%) (Per-Protocol Population)
Description: Summary statistics of percent change from Baseline for urinary S-phenyl mercapturic acid [S-PMA] (%) in each study visit are presented.
  Baseline taken from Visit 3 (Day 8±1) value. Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
  Mean percent change from baseline is the mean of all individual subjects' percent change from baseline values. Each percent change from baseline was calculated by subtracting the individual subject's baseline value from the value at the desired timepoint and then dividing this calculated value by the individual subject's baseline value and multiplying by 100. These individual subjects' percent changes from baseline values were used to calculate the mean percent change from baseline using a SAS® procedure.
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
percent change from baseline
  Visit 4: number analyzed (Participants) | 79 | 50
  Visit 4 | 17.5 (67.39) | 21.1 (77.37)
  Visit 5: number analyzed (Participants) | 82 | 49
  Visit 5 | 13.4 (67.41) | 38.2 (69.68)
  Visit 6: number analyzed (Participants) | 74 | 51
  Visit 6 | 19.7 (60.60) | 44.4 (87.87)
  End of Study/Early Termination: number analyzed (Participants) | 81 | 51
  End of Study/Early Termination | 20.9 (76.27) | 39.1 (70.93)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study in S-PMA; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study in S-PMA; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study in S-PMA; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study in S-PMA; p = 0.1524, t-test, 2 sided; Mean Difference (Net) = -19.0, 95% CI 2-sided [-45.1 to 7.12] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 6, analysis 1]; Test type: Equivalence — [test comment as in outcome 6, analysis 1]; p = 0.4014, t-test, 2 sided; Mean Difference (Net) = -12.1, 95% CI 2-sided [-40.4 to 16.3] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Summary Statistics of Change From Baseline for Carboxyhemoglobin (%) (Per-Protocol Population)
Description: Summary statistics of change from Baseline for blood carboxyhemoglobin (%) in each study visit are presented.
  Baseline taken from Visit 3 (Day 8±1) value. Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: percent saturation of carboxyhemoglobin
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
percent saturation of carboxyhemoglobin
  Visit 4 | -0.42 (1.449) | 0.03 (1.460)
  Visit 5: number analyzed (Participants) | 86 | 55
  Visit 5 | -0.24 (1.418) | 0.39 (1.374)
  Visit 6 | -0.02 (1.547) | 0.39 (1.299)
  End of Study/Early Termination | -0.61 (1.387) | -0.10 (1.118)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in carboxyhemoglobin; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in carboxyhemoglobin; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in carboxyhemoglobin; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in carboxyhemoglobin; p = 0.0241, t-test, 2 sided; Mean Difference (Net) = -0.507, 95% CI 2-sided [-0.946 to -0.0674] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 7, analysis 1]; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p = 0.1292, t-test, 2 sided; Mean Difference (Net) = -0.367, 95% CI 2-sided [-0.843 to 0.108] — [estimate comment as in outcome 2, analysis 2]

8. Secondary Outcome: Summary Statistics of Percent Change From Baseline for Carboxyhemoglobin (%) (Per-Protocol Population)
Description: Summary statistics of percent change from Baseline for blood carboxyhemoglobin (%) in each study visit are presented.
  Baseline taken from Visit 3 (Day 8±1) value. Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
  Mean percent change from baseline is the mean of all individual subjects' percent change from baseline values. Each percent change from baseline was calculated by subtracting the individual subject's baseline value from the value at the desired timepoint and then dividing this calculated value by the individual subject's baseline value and multiplying by 100. These individual subjects' percent changes from baseline values were used to calculate the mean percent change from baseline using a SAS® procedure.
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
percent change from baseline
  Visit 4 | -6.3 (27.48) | 5.3 (35.59)
  Visit 5: number analyzed (Participants) | 86 | 55
  Visit 5 | -4.0 (26.17) | 9.8 (27.21)
  Visit 6 | 1.4 (28.26) | 11.3 (29.44)
  End of Study/Early Termination | -9.3 (27.89) | 0.7 (25.53)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study in carboxyhemoglobin; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study in carboxyhemoglobin; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study in carboxyhemoglobin; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study in carboxyhemoglobin; p = 0.0333, t-test, 2 sided; Mean Difference (Net) = -10.0, 95% CI 2-sided [-19.2 to -0.803] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 8, analysis 1]; Test type: Equivalence — [test comment as in outcome 8, analysis 1]; p = 0.1767, t-test, 2 sided; Mean Difference (Net) = -6.76, 95% CI 2-sided [-16.6 to 3.08] — [estimate comment as in outcome 1, analysis 2]

9. Secondary Outcome: Summary Statistics of Change From Baseline for Exhaled Carbon Monoxide (Ppm) (Per-Protocol Population)
Description: Summary statistics of change from Baseline for exhaled carbon monoxide (ppm) in each study visit are presented.
  Baseline taken from Visit 3 (Day 8±1) value. Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
ppm
  Visit 4 | -1.4 (9.41) | -0.2 (7.84)
  Visit 5 | -1.9 (7.48) | 0.7 (8.37)
  Visit 6 | -0.8 (9.30) | 0.6 (7.89)
  End of Study/Early Termination | -2.3 (9.17) | -0.8 (6.90)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in exhaled carbon monoxide; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in exhaled carbon monoxide; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in exhaled carbon monoxide; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in exhaled carbon monoxide; p = 0.2961, t-test, 2 sided; Mean Difference (Net) = -1.51, 95% CI 2-sided [-4.36 to 1.34] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 9, analysis 1]; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; p = 0.5015, t-test, 2 sided; Mean Difference (Net) = -1.05, 95% CI 2-sided [-4.12 to 2.03] — [estimate comment as in outcome 2, analysis 2]

10. Secondary Outcome: Summary Statistics of Percent Change From Baseline for Exhaled Carbon Monoxide (%) (Per-Protocol Population)
Description: Summary statistics of percent change from Baseline for exhaled carbon monoxide (%) in each study visit are presented.
  Baseline taken from Visit 3 (Day 8±1) value. Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
  Mean percent change from baseline is the mean of all individual subjects' percent change from baseline values. Each percent change from baseline was calculated by subtracting the individual subject's baseline value from the value at the desired timepoint and then dividing this calculated value by the individual subject's baseline value and multiplying by 100. These individual subjects' percent changes from baseline values were used to calculate the mean percent change from baseline using a SAS® procedure.
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
percent change from baseline
  Visit 4 | -0.8 (44.65) | 12.0 (65.86)
  Visit 5 | -5.8 (37.05) | 11.4 (54.87)
  Visit 6 | 3.5 (49.07) | 13.9 (57.42)
  End of Study/Early Termination | -3.1 (47.00) | 9.0 (66.04)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study in exhaled carbon monoxide; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study in exhaled carbon monoxide; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study in exhaled carbon monoxide; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study in exhaled carbon monoxide; p = 0.2048, t-test, 2 sided; Mean Difference (Net) = -12.1, 95% CI 2-sided [-30.9 to 6.68] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to control in exhaled carbon monoxide; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to control in exhaled carbon monoxide; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to control in exhaled carbon monoxide; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to control in exhaled carbon monoxide; p = 0.4731, t-test, 2 sided; Mean Difference (Net) = -7.32, 95% CI 2-sided [-27.4 to 12.8] — [estimate comment as in outcome 1, analysis 2]

11. Secondary Outcome: Summary Statistics of Change From Baseline in Cigarettes Smoked Per Day (Per-Protocol Population)
Description: Summary statistics of change from Baseline in number or products used day in each study visit are presented.
  Values for visit are the average of daily values for the previous week Visit 4 = Day 15±1 Visit 5 = Day 22±1 Visit 6 = Day 29±1 Visit 7/End of Study = Day 36±1
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
cigarettes per day
  Visit 4 | -2.7 (3.28) | 0.5 (1.96)
  Visit 5 | -3.1 (4.34) | 0.3 (2.37)
  Visit 6 | -2.9 (4.41) | 0.3 (2.78)
  End of Study/Early Termination: number analyzed (Participants) | 85 | 55
  End of Study/Early Termination | -3.5 (4.78) | 0.4 (2.76)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in cigarettes smoked per day; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in cigarettes smoked per day; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of change from baseline in cigarettes smoked per day; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline in cigarettes smoked per day; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = -3.86, 95% CI 2-sided [-5.25 to -2.47] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 11, analysis 1]; Test type: Equivalence — [test comment as in outcome 11, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = -3.74, 95% CI 2-sided [-5.14 to -2.34] — [estimate comment as in outcome 2, analysis 2]

12. Secondary Outcome: Summary Statistics of Percent Change From Baseline for Cigarettes Smoked Per Day (CPD) (Per-Protocol Population)
Description: Summary statistics of percent change from Baseline of number of products used per day in each study visit are presented.
  CPD was tracked using an interactive voice response system (IVRS). During the Baseline Period (Days 1 to 8), subjects reported CPD daily through an IVRS each day between 16:00 and 19:00. Test and Control subjects continued daily tobacco use tracking via an IVRS and return to the study site once a week during the 4 week Product Use Period on Days 15, 22, 29, and 36.
  Mean percent change from baseline is the mean of all individual subjects' percent change from baseline values. Each percent change from baseline was calculated by subtracting the individual subject's baseline value from the value at the desired timepoint and then dividing the calculated value by the individual subject's baseline value and multiplying by 100. These individual subjects' percent changes from baseline values were used to calculate the mean percent change from baseline using a SAS procedure.
Time Frame: as for outcome 1
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
percent change from baseline
  Visit 4 | -15.0 (19.30) | 3.1 (10.85)
  Visit 5 | -16.5 (26.21) | 2.9 (15.18)
  Visit 6 | -16.3 (24.78) | 2.9 (18.01)
  End of Study/Early Termination: number analyzed (Participants) | 85 | 55
  End of Study/Early Termination | -19.2 (27.03) | 3.2 (17.28)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study in cigarettes smoked per day; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study in cigarettes smoked per day; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study in cigarettes smoked per day; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study in cigarettes smoked per day; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = -22.5, 95% CI 2-sided [-30.5 to -14.5] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 12, analysis 1]; Test type: Equivalence — [test comment as in outcome 12, analysis 1]; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = -22.3, 95% CI 2-sided [-30.4 to -14.1] — [estimate comment as in outcome 1, analysis 2]

13. Secondary Outcome: Summary Statistics of Change From Baseline for Total Score of Fagerstrom Test for Cigarette Dependence (Per-Protocol Population)
Description: Summary statistics of change from Baseline for Total Score of Fagerstrom Test for Cigarette Dependence at the end of study/early termination are presented. The Fagerstrom Test for Nicotine Dependence consists of Yes/No and multiple-choice questions where each response is assigned a value from 0 to 1 (for yes/no questions) or 0 to 3 (for multiple-choice questions). Values are summed to yield a total score with a minimum score of 0 points and a maximum score of 10 points. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
  Baseline = Visit 3 (Day 8) value Population: Per-Protocol
Time Frame: Day 36 (Visit 7/End of Study) relative to the start of the baseline period (Visit 2/Day 1)
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 86 | 55
scores on a scale | -0.4 (1.66) | 0.0 (0.82)
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of change from baseline to end of study for Fagerstrom Test score for Cigarette Dependence; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline to end of study for Fagerstrom Test score for Cigarette Dependence; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of change from baseline to end of study for Fagerstrom Test score for Cigarette Dependence; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change from baseline to end of study for Fagerstrom Test score for Cigarette Dependence; p = 0.0919, t-test, 2 sided; Mean Difference (Net) = -0.408, 95% CI 2-sided [-0.884 to 0.0673] — Difference in LS mean change between study groups using Mixed Effects Repeated Measures Model 1: Change from baseline=study group + visit + study group*visit + subject + random error, fitted with unstructured covariance matrix
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 13, analysis 1]; Test type: Equivalence — [test comment as in outcome 13, analysis 1]; p = 0.0975, t-test, 2 sided; Mean Difference (Net) = -0.405, 95% CI 2-sided [-0.886 to 0.0751] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Statistical Analysis of Difference in Percent Change from Baseline in Total Score of Fagerstrom Test for Cigarette Dependence between the Study Groups. Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study for Fagerstrom Test score for Cigarette Dependence; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study for Fagerstrom Test score for Cigarette Dependence; Test type: Equivalence — Statistical Analysis of Difference in Percent Change from Baseline in Total Score of Fagerstrom Test for Cigarette Dependence between the Study Groups. Null hypothesis = Test and Control groups will have equivalent levels of percent change from baseline to end of study for Fagerstrom Test score for Cigarette Dependence; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of percent change from baseline to end of study for Fagerstrom Test score for Cigarette Dependence; p = 0.0643, t-test, 2 sided; Mean Difference (Net) = -8.31, 95% CI 2-sided [-17.1 to 0.499] — Difference in LS mean percent change between study groups using Mixed Effects Repeated Measures Model 1: Change from baseline=study group + visit + study group*visit + subject + random error, fitted with unstructured covariance matrix
Statistical Analysis 4: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 13, analysis 3]; Test type: Equivalence — [test comment as in outcome 13, analysis 3]; p = 0.0517, t-test, 2 sided; Mean Difference (Net) = -8.84, 95% CI 2-sided [-17.7 to 0.0661] — [estimate comment as in outcome 2, analysis 2]

14. Secondary Outcome: Count of Subjects in Subgroups Based on Change From Baseline to End of Study on Change in Quit Attempts (Per-Protocol)
Description: Count of Test and Control subjects that reported an increase, decrease or no change in quit attempts from Baseline to End of Study are presented. Results for the number of self-reported attempts to quit smoking in the previous 30 days were collected from subject responses to the question "How many times during the past 30 days have you stopped smoking cigarettes for 24 hours or longer because you were trying to quit?".
  Baseline = Visit 2 values. Population: Per-Protocol.
Time Frame: Day 36 (Visit 7/End of Study) relative to the start of the baseline period (Visit 2/Day 1)
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 87 | 55
Participants
  Increase | 4 | 0
  No Change | 82 | 53
  Decrease | 1 | 2
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of change in quit attempts from baseline to end of study; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change in quit attempts from baseline to end of study; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of change in quit attempts from baseline to end of study; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change in quit attempts from baseline to end of study; p = 0.2160, Fisher Exact; Probability = 0.2160 — Estimated value is the probability of observed distribution assuming the null hypothesis
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 14, analysis 1]; Test type: Equivalence — [test comment as in outcome 14, analysis 1]; p = 0.0648, Cochran-Mantel-Haenszel; Probability = 0.0648

15. Secondary Outcome: Count of Subjects in Subgroups Based on Change From Baseline to End of Study on Change in Quitting Intentions (Per-Protocol)
Description: Count of Test and Control subjects that reported a change (No to Yes) or no change in quitting intentions from Baseline to End of Study are presented. Results were collected from subject Yes/No responses to the question "Are you planning to quit smoking in the next 30 days?".
  Baseline = Visit 2 responses. Population: Per-Protocol.
Time Frame: Day 36 (Visit 7/End of Study) relative to the start of the baseline period (Visit 2/Day 1)
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 86 | 50
Participants
  No to Yes | 12 | 5
  Same | 74 | 45
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent levels of change in quitting intentions from baseline to end of study; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change in quitting intentions from baseline to end of study; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent levels of change in quitting intentions from baseline to end of study; Alternate hypothesis = Test and Control groups will NOT have equivalent levels of change in quitting intentions from baseline to end of study; p = 0.5977, Fisher Exact; Probability = 0.5977 — Estimated value is the probability of observed distribution assuming the null hypothesis

16. Secondary Outcome: Difference in Means of Urinary Total NNAL Exposure Between Day 1 and Day 8 (Per-Protocol)
Description: This secondary objective was to compare differences in the biomarker of exposure between two methods for determining CPD during the Baseline Period.
  Difference in mean urinary total NNAL exposure between two methods for determining daily product use (Cigarettes Per Day [CPD]) during the Baseline Period:
  Method 1: Recall of average daily CPD for prior week using Past 7 Day Cigarettes Use Questionnaire (Day 1).
  Method 2: Daily CPD tracking using an interactive voice response system (IVRS; 7 day average of values recorded on Days 2 through 8).
  Population: Per-Protocol.
Time Frame: Daily during Baseline Period (Day 1 to Day 8)
Population: The CPD from Method 1 (Past 7 Day Cigarettes Use Questionnaire) for all subjects in the Per-Protocol population was compared to CPD from Method 2 (7 day average from IVRS) for all subjects in the Per-Protocol population.
Measure: Mean (Standard Deviation); unit: ng/g
Groups:
- Day 1 (Weekly Recall): Recall of average daily CPD for prior week using Past 7 Day Cigarettes Use Questionnaire (Day 1)
- Day 8 (Daily Tracking Using IVRS): Daily CPD tracking using an interactive voice response system (IVRS; 7 day average of values recorded on Days 2 through 8).
Arm/Group | Day 1 (Weekly Recall) | Day 8 (Daily Tracking Using IVRS)
Number analyzed (Participants) | 138 | 138
ng/g | 485.0 (348.45) | 495.0 (358.54)
Statistical Analysis 1: Comparison: Day 1 (Weekly Recall) vs Day 8 (Daily Tracking Using IVRS); Null hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will have equivalent levels of change in mean exposure of NNAL; Alternate hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT have equivalent levels of change from baseline to end of study in mean exposure of NNAL; Test type: Equivalence — Null hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will have equivalent levels of change in mean exposure of NNAL; Alternate hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT have equivalent levels of change from baseline to end of study in mean exposure of NNAL; p = 0.4388, t-test, 2 sided; Mean Difference (Net) = 10.0, 95% CI 2-sided [-15.5 to 35.5]

17. Secondary Outcome: Difference in Means of Nicotine Equivalents Exposure Between Day 1 and Day 8 (Per-Protocol)
Description: This secondary objective was to compare differences in the biomarker of exposure between two methods for determining CPD during the Baseline Period.
  Difference in mean urinary nicotine equivalents exposure between two methods for determining daily product use (Cigarettes Per Day [CPD]) during the Baseline Period:
  Method 1: Recall of average daily CPD for prior week using Past 7 Day Cigarettes Use Questionnaire (Day 1).
  Method 2: Daily CPD tracking using an interactive voice response system (IVRS; 7 day average of values recorded on Days 2 through 8).
  Nicotine equivalents include nicotine and its 5 metabolites (cotinine, trans-3'-hydroxycotinine, trans-3'-hydroxycotinine-0-glucuronide, nicotine-N-glucuronide, and cotinine-N-glucuronide) Population: Per-Protocol.
Time Frame: Daily during Baseline Period (Day 1 to Day 8)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Day 1 (Weekly Recall) | Day 8 (Daily Tracking Using IVRS)
Number analyzed (Participants) | 122 | 122
mg/g | 13.29 (9.138) | 13.74 (9.049)
Statistical Analysis 1: Comparison: Day 1 (Weekly Recall) vs Day 8 (Daily Tracking Using IVRS); Null hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will have equivalent levels of change in mean exposure of nicotine metabolites; Alternate hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT have equivalent levels of change from baseline to end of study in mean exposure of nicotine metabolites; Test type: Equivalence — Null hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will have equivalent levels of change in mean exposure of nicotine metabolites; Alternate hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT have equivalent levels of change from baseline to end of study in mean exposure of nicotine metabolites; p = 0.3390, t-test, 2 sided; Mean Difference (Net) = 0.45, 95% CI 2-sided [-0.48 to 1.38]

18. Secondary Outcome: Difference in Means of S-PMA Exposure Between Day 1 and Day 8 (Per-Protocol)
Description: This secondary objective was to compare differences in the biomarker of exposure between two methods for determining CPD during the Baseline Period.
  Difference in mean urinary S-phenylmercapturic acid [S-PMA] exposure between two methods for determining daily product use (Cigarettes Per Day [CPD]) during the Baseline Period:
  Method 1: Recall of average daily CPD for prior week using Past 7 Day Cigarettes Use Questionnaire (Day 1).
  Method 2: Daily CPD tracking using an interactive voice response system (IVRS; 7 day average of values recorded on Days 2 through 8).
  Population: Per-Protocol.
Time Frame: Daily during Baseline Period (Day 1 to Day 8)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Day 1 (Weekly Recall) | Day 8 (Daily Tracking Using IVRS)
Number analyzed (Participants) | 136 | 136
ng/g | 5773 (5786.3) | 5567 (5222.3)
Statistical Analysis 1: Comparison: Day 1 (Weekly Recall) vs Day 8 (Daily Tracking Using IVRS); Null hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will have equivalent levels of change in mean exposure of S-PMA; Alternate hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT have equivalent levels of change from baseline to end of study in mean exposure of S-PMA; Test type: Equivalence — Null hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will have equivalent levels of change in mean exposure of S-PMA; Alternate hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT have equivalent levels of change from baseline to end of study in mean exposure of S-PMA; p = 0.4526, t-test, 2 sided; Mean Difference (Net) = -205, 95% CI 2-sided [-745 to 334]

19. Secondary Outcome: Difference in Means of Carboxyhemoglobin (COHb) Exposure Between Day 1 and Day 8 (Per-Protocol)
Description: This secondary objective was to compare differences in the biomarker of exposure between two methods for determining CPD during the Baseline Period.
  Difference in mean blood carboxyhemoglobin [COHb] exposure between two methods for determining daily product use (Cigarettes Per Day [CPD]) during the Baseline Period:
  Method 1: Recall of average daily CPD for prior week using Past 7 Day Cigarettes Use Questionnaire (Day 1).
  Method 2: Daily CPD tracking using an interactive voice response system (IVRS; 7 day average of values recorded on Days 2 through 8).
  Population: Per-Protocol.
Time Frame: Daily during Baseline Period (Day 1 to Day 8)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percent saturation of carboxyhemoglobin
Arm/Group | Day 1 (Weekly Recall) | Day 8 (Daily Tracking Using IVRS)
Number analyzed (Participants) | 142 | 142
percent saturation of carboxyhemoglobin | 5.4 (2.13) | 5.4 (1.96)
Statistical Analysis 1: Comparison: Day 1 (Weekly Recall) vs Day 8 (Daily Tracking Using IVRS); Null hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will have equivalent levels of change in mean exposure of carboxyhemoglobin; Alternate hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT have equivalent levels of change from baseline to end of study in mean exposure of carboxyhemoglobin; Test type: Equivalence — Null hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will have equivalent levels of change in mean exposure of carboxyhemoglobin; Alternate hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT have equivalent levels of change from baseline to end of study in mean exposure of carboxyhemoglobin; p = 0.9440, t-test, 2 sided; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

20. Secondary Outcome: Difference in Means of Carbon Monoxide (CO) Exposure Between Day 1 and Day 8 (Per-Protocol)
Description: This secondary objective was to compare differences in the biomarker of exposure between two methods for determining CPD during the Baseline Period.
  Difference in mean exhaled carbon monoxide [CO] between two methods for determining daily product use (Cigarettes Per Day, CPD) during the Baseline Period:
  Method 1: Recall of average daily CPD for prior week using Past 7 Day Cigarettes Use Questionnaire (Day 1).
  Method 2: Daily CPD tracking using an interactive voice response system (IVRS; 7 day average of values recorded on Days 2 through 8).
  Population: Per-Protocol.
Time Frame: Daily during Baseline Period (Day 1 to Day 8)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Day 1 (Weekly Recall) | Day 8 (Daily Tracking Using IVRS)
Number analyzed (Participants) | 142 | 142
ppm | 22 (10.0) | 22 (10.3)
Statistical Analysis 1: Comparison: Day 1 (Weekly Recall) vs Day 8 (Daily Tracking Using IVRS); Null hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will have equivalent levels of change in mean exposure of carbon monoxide; Alternate hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT have equivalent levels of change from baseline to end of study in mean exposure of carbon monoxide; Test type: Equivalence — Null hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will have equivalent levels of change in mean exposure of carbon monoxide; Alternate hypothesis = The Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT have equivalent levels of change from baseline to end of study in mean exposure of carbon monoxide; p = 0.7484, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [-1 to 1]

21. Secondary Outcome: Difference in Cigarettes Per Day Between the Once Weekly Recall at Day 8 (From Questionnaire) and the Average Daily Tracking Days 2 Through 8 (From IVRS) (Per-Protocol)
Description: This secondary objective was to compare differences in the biomarker of exposure between two methods for determining CPD during the Baseline Period.
  Difference in product use (Cigarettes Per Day [CPD]), including test product, between two methods for determining CPD during the Baseline Period:
  Method 1: Recall of average daily CPD for prior week using Past 7 Day Cigarettes Use Questionnaire (Day 1).
  Method 2: Daily CPD tracking using an interactive voice response system (IVRS; 7 day average of values recorded on Days 2 through 8).
  Population: Per-Protocol.
Time Frame: Daily during Baseline Period (Day 1 to Day 8)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Day 1 (Weekly Recall) | Day 8 (Daily Tracking Using IVRS)
Number analyzed (Participants) | 129 | 129
cigarettes per day | 19 (6.4) | 19 (6.3)
Statistical Analysis 1: Comparison: Day 1 (Weekly Recall) vs Day 8 (Daily Tracking Using IVRS); Null hypothesis = Cigarette consumption (CPD) determined using the Day 1 (Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will be equivalent; Alternate hypothesis = Cigarette consumption (CPD) determined using the Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT be equivalent; Test type: Equivalence — Null hypothesis = Cigarette consumption (CPD) determined using the Day 1 (Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will be equivalent; Alternate hypothesis = Cigarette consumption (CPD) determined using the Day 1(Weekly Recall) and Day 8 (Daily Tracking using IVRS) methods will NOT be equivalent; p = 0.9992, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [0 to 0]

22. Secondary Outcome: Frequency and Percentage of Subjects With Change From Baseline in Cigarette Consumption
Description: Change in cigarette consumption, categorized as 'No change', '<50% reduction', '50% to < 100% reduction', '100% reduction' or 'Increase', among subjects in Test and Control groups are presented. Baseline values are based on the average of daily values for the week prior to randomization (Visit 3/Day 8±1).
Time Frame: Day 15 (Visit 4), Day 22 (Visit 5), Day 29 (Visit 6) and Day 36 (Visit 7)
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Groups:
- Test (Visit 4): Change in Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) cigarette consumption from Baseline to Visit 4
- Control (Visit 4): Change in Control Group (subjects continued ad libitum use of their own brand of tobacco products) cigarette consumption from Baseline to Visit 4
- Test (Visit 5): Change in Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) cigarette consumption from Baseline to Visit 5
- Control (Visit 5): Change in Control Group (subjects continued ad libitum use of their own brand of tobacco products) cigarette consumption from Baseline to Visit 5
- Test (Visit 6): Change in Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) cigarette consumption from Baseline to Visit 6
- Control (Visit 6): Change in Control Group (subjects continued ad libitum use of their own brand of tobacco products) cigarette consumption from Baseline to Visit 6
- Test (End of Study): Change in Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) cigarette consumption from Baseline to End of Study
- Control (End of Study): Change in Control Group (subjects continued ad libitum use of their own brand of tobacco products) cigarette consumption from Baseline to End of Study
Arm/Group | Test (Visit 4) | Control (Visit 4) | Test (Visit 5) | Control (Visit 5) | Test (Visit 6) | Control (Visit 6) | Test (End of Study) | Control (End of Study)
Number analyzed (Participants) | 87 | 55 | 87 | 55 | 87 | 55 | 85 | 55
Participants
  No Change | 5 | 3 | 6 | 4 | 6 | 4 | 8 | 2
  <50% Reduction | 67 | 22 | 62 | 21 | 56 | 25 | 57 | 24
  50% to < 100% | 3 | 0 | 3 | 0 | 7 | 0 | 8 | 0
  100% Reduction | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0
  Increase | 12 | 30 | 14 | 30 | 17 | 26 | 10 | 29

23. Secondary Outcome: Frequency and Percentage of Subjects With Change From Baseline in Urinary Total NNAL (ng / g Creatinine)
Description: Change in Urinary Total NNAL, categorized as 'No change', 'Reduction', 'Increase' or 'Missing', among subjects in Test and Control groups are presented. Baseline values are Visit 3 (Day 8) values.
Time Frame: Day 15 (Visit 4), Day 22 (Visit 5), Day 29 (Visit 6) and Day 36 (Visit 7)
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Groups:
- Control (Visit 4): Change in Control Group cigarette (subjects continued ad libitum use of their own brand of tobacco products) consumption from Baseline to Visit 4
- Control (Visit 5): Change in Control Group cigarette (subjects continued ad libitum use of their own brand of tobacco products) consumption from Baseline to Visit 5
- Control (Visit 6): Change in Control Group cigarette (subjects continued ad libitum use of their own brand of tobacco products) consumption from Baseline to Visit 6
- Control (End of Study): Change in Control Group cigarette (subjects continued ad libitum use of their own brand of tobacco products) consumption from Baseline to End of Study
Arm/Group | Test (Visit 4) | Control (Visit 4) | Test (Visit 5) | Control (Visit 5) | Test (Visit 6) | Control (Visit 6) | Test (End of Study) | Control (End of Study)
Number analyzed (Participants) | 87 | 55 | 87 | 55 | 87 | 55 | 87 | 55
Participants
  No Change | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reduction | 45 | 25 | 40 | 18 | 33 | 16 | 38 | 18
  Increase | 35 | 28 | 43 | 33 | 46 | 37 | 46 | 36
  Missing | 7 | 2 | 4 | 4 | 8 | 2 | 3 | 1

24. Secondary Outcome: Frequency and Percentage of Subjects With Change From Baseline in Quitting Intentions
Description: Change in subject quitting intentions from Baseline to End of Study are presented. Subject responses were categorized as 'No to Yes', 'Yes to No' and 'Same' (no change in quitting intention). Baseline = Visit 2 (Day 1)
Time Frame: Day 36 (Visit 7/End of Study) relative to the start of the baseline period (Visit 2/Day 1)
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Groups:
- Test: Subjects were allowed to continue smoking their own brand of cigarettes ad libitum and were provided the option to use the test product (VBM-FG2 oral discs) also under ad libitum conditions
- Control: Subjects continued ad libitum use of their own brand of cigarettes and/or other tobacco products throughout the study but were not provided the test product (VBM-FG2 oral discs) for use in the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 86 | 50
Participants
  No to Yes | 12 | 5
  Yes to No | 0 | 0
  Same | 74 | 45

25. Secondary Outcome: Summary Statistics of Cigarettes Smoked Per Day on Visits 2 (Day 1) and 3 (Day 8)
Description: Summary statistics of average cigarettes smoked per day [CPD] over previous 7 days collected from Cigarette Use questionnaire on Visit 2 (Day 1) and Visit 3 (Day 8) are presented.
Time Frame: Day 1 (Visit 2) and Day 8 (Visit 3)
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: cigarettes per day
Groups:
- Test (Visit 2): Summary statistics of CPD for Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) on Visit 2
- Control (Visit 2): Summary statistics of CPD for Control Group (subjects continued ad libitum use of their own brand of tobacco products) on Visit 2
- Test (Visit 3): Summary statistics of CPD for Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) on Visit 3
- Control (Visit 3): Summary statistics of CPD for Control Group (subjects continued ad libitum use of their own brand of tobacco products) on Visit 3
Arm/Group | Test (Visit 2) | Control (Visit 2) | Test (Visit 3) | Control (Visit 3)
Number analyzed (Participants) | 74 | 50 | 79 | 50
cigarettes per day | 17.7 (6.04) | 19.8 (7.64) | 17.6 (5.36) | 20.0 (7.43)

26. Secondary Outcome: Summary Statistics of Carboxyhemoglobin by Study Group and Cigarette Consumption Categories Over Visits
Description: Summary statistics of blood carboxyhemoglobin in each visit among subjects in Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
Time Frame: Day 1 (Visit 2), Day 8 (Visit 3), Day 15 (Visit 4), Day 22 (Visit 5), Day 29 (Visit 6) and Day 36 (Visit 7)
Population: The CPD frequency population (the subjects from the per-protocol population in each cigarette consumption category) was defined by the end of study cigarette use data. This population was then assessed for biomarker data at end of study and previous study visits. The number of samples for biomarkers data may not equal the number of subjects in population (defined by end of study CPD), due to missing visits, missing samples, or missing analytical results.
Measure: Mean (Standard Deviation); unit: percent saturation of carboxyhemoglobin
Groups:
- Test (Visit 2): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Visit 2
- Control (Visit 2): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Visit 2
- Test (Visit 3): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Visit 3
- Control (Visit 3): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Visit 3
- Test (Visit 4): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Visit 4
- Control (Visit 4): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Visit 4
- Test (Visit 5): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Visit 5
- Control (Visit 5): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Visit 5
- Test (Visit 6): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Visit 6
- Control (Visit 6): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Visit 6
- Test (End of Study): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) End of Study
- Control (End of Study): Control Group (subjects continued ad libitum use of their own brand of tobacco products) End of Study
Arm/Group | Test (Visit 2) | Control (Visit 2) | Test (Visit 3) | Control (Visit 3) | Test (Visit 4) | Control (Visit 4) | Test (Visit 5) | Control (Visit 5) | Test (Visit 6) | Control (Visit 6) | Test (End of Study) | Control (End of Study)
Number analyzed (Participants) | 87 | 55 | 87 | 55 | 87 | 55 | 86 | 55 | 87 | 55 | 87 | 55
percent saturation of carboxyhemoglobin
  Increase: number analyzed (Participants) | 11 | 29 | 11 | 29 | 11 | 29 | 11 | 29 | 11 | 29 | 11 | 29
  Increase | 6.5 (2.61) | 5.5 (2.10) | 6.6 (2.15) | 5.3 (1.63) | 6.2 (2.15) | 5.5 (1.65) | 6.8 (2.46) | 6.1 (2.26) | 6.6 (2.15) | 5.8 (2.07) | 6.0 (1.80) | 5.4 (1.79)
  No Change: number analyzed (Participants) | 8 | 2 | 8 | 2 | 8 | 2 | 8 | 2 | 8 | 2 | 8 | 2
  No Change | 4.7 (1.57) | 3.9 (0.14) | 5.7 (2.15) | 3.7 (2.19) | 5.2 (1.73) | 3.3 (0.14) | 5.2 (1.76) | 3.2 (0.07) | 4.9 (1.42) | 5.6 (3.11) | 5.0 (1.28) | 4.6 (1.41)
  <50% Reduction: number analyzed (Participants) | 56 | 24 | 56 | 24 | 56 | 24 | 55 | 24 | 56 | 24 | 56 | 24
  <50% Reduction | 5.5 (2.01) | 5.0 (2.35) | 5.4 (1.92) | 5.0 (2.18) | 5.2 (2.05) | 4.8 (2.15) | 5.4 (2.24) | 5.0 (2.08) | 5.8 (2.28) | 5.1 (1.82) | 5.1 (2.07) | 4.6 (1.85)
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 0 | 8 | 0 | 8 | 0 | 8 | 0
  50% to < 100% Reduction | 5.0 (2.5) |  | 5.4 (2.16) |  | 4.7 (2.03) |  | 4.4 (1.98) |  | 3.7 (1.90) |  | 3.2 (1.87) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 4.5 (0.14) |  | 4.5 (0.35) |  | 2.0 (0.64) |  | 1.2 (0.21) |  | 1.2 (0.00) |  | 1.5 (0.21) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 3.5 (1.63) |  | 4.3 (2.33) |  | 2.2 (0.14) |  | 3.3 (1.98) |  | 4.1 (1.91) |  | 3.7 (0.92) |
  Overall | 5.4 (2.11) | 5.3 (2.18) | 5.5 (1.99) | 5.1 (1.90) | 5.1 (2.10) | 5.1 (1.91) | 5.3 (2.32) | 5.5 (2.23) | 5.5 (2.33) | 5.5 (1.98) | 4.9 (2.07) | 5.0 (1.82)

27. Secondary Outcome: Summary Statistics of Exhaled Carbon Monoxide by Study Group and Cigarette Consumption Categories Over Visits
Description: Summary Statistics of exhaled carbon monoxide in each visit among subjects in Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
Time Frame: Day 1 (Visit 2), Day 8 (Visit 3), Day 15 (Visit 4), Day 22 (Visit 5), Day 29 (Visit 6) and Day 36 (Visit 7)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Test (Visit 2) | Control (Visit 2) | Test (Visit 3) | Control (Visit 3) | Test (Visit 4) | Control (Visit 4) | Test (Visit 5) | Control (Visit 5) | Test (Visit 6) | Control (Visit 6) | Test (End of Study) | Control (End of Study)
Number analyzed (Participants) | 87 | 55 | 87 | 55 | 87 | 55 | 87 | 55 | 87 | 55 | 87 | 55
ppm
  Increase: number analyzed (Participants) | 11 | 29 | 11 | 29 | 11 | 29 | 11 | 29 | 11 | 29 | 11 | 29
  Increase | 28.3 (11.13) | 21.0 (9.65) | 29.6 (12.12) | 20.6 (9.11) | 28.5 (15.29) | 21.4 (8.57) | 28.1 (13.60) | 22.7 (13.28) | 27.8 (12.32) | 21.8 (10.44) | 25.9 (8.86) | 20.2 (9.54)
  No Change: number analyzed (Participants) | 8 | 2 | 8 | 2 | 8 | 2 | 8 | 2 | 8 | 2 | 8 | 2
  No Change | 17.3 (10.77) | 15.5 (3.54) | 22.5 (9.56) | 11.5 (10.61) | 21.6 (8.88) | 12.0 (4.24) | 22.4 (10.88) | 11.5 (2.12) | 19.3 (9.82) | 18.0 (9.90) | 21.5 (9.96) | 18.5 (2.12)
  <50% Reduction: number analyzed (Participants) | 56 | 24 | 56 | 24 | 56 | 24 | 56 | 24 | 56 | 24 | 56 | 24
  <50% Reduction | 22.2 (9.21) | 22.3 (10.87) | 21.6 (10.01) | 21.0 (11.13) | 20.9 (11.16) | 19.4 (10.89) | 20.5 (10.25) | 19.9 (9.98) | 23.0 (11.32) | 20.4 (9.24) | 21.1 (10.09) | 19.1 (8.71)
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 0 | 8 | 0 | 8 | 0 | 8 | 0
  50% to < 100% Reduction | 19.3 (12.14) |  | 20.6 (9.86) |  | 18.0 (8.83) |  | 15.5 (8.38) |  | 12.1 (8.54) |  | 9.9 (6.08) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 20.0 (5.66) |  | 17.0 (4.24) |  | 4.5 (0.71) |  | 2.5 (0.71) |  | 5.5 (2.12) |  | 4.0 (2.83) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 20.5 (14.85) |  | 18.5 (16.26) |  | 10.5 (2.12) |  | 9.5 (6.36) |  | 15.5 (12.02) |  | 13.0 (8.49) |
  Overall | 22.1 (10.05) | 21.4 (10.03) | 22.4 (10.40) | 20.4 (10.05) | 21.0 (11.68) | 20.2 (9.62) | 20.5 (11.18) | 21.1 (11.81) | 21.7 (11.71) | 21.0 (9.77) | 20.1 (10.41) | 19.7 (8.94)

28. Secondary Outcome: Summary Statistics of S-PMA by Study Group and Cigarette Consumption Categories Over Visits
Description: Summary statistics of urinary S-PMA (ng/g creatinine) in each visit among subjects in Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
Time Frame: Day 1 (Visit 2), Day 8 (Visit 3), Day 15 (Visit 4), Day 22 (Visit 5), Day 29 (Visit 6) and Day 36 (Visit 7)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test (Visit 2) | Control (Visit 2) | Test (Visit 3) | Control (Visit 3) | Test (Visit 4) | Control (Visit 4) | Test (Visit 5) | Control (Visit 5) | Test (Visit 6) | Control (Visit 6) | Test (End of Study) | Control (End of Study)
Number analyzed (Participants) | 85 | 54 | 84 | 54 | 80 | 50 | 84 | 49 | 77 | 52 | 83 | 52
ng/g
  Increase: number analyzed (Participants) | 11 | 28 | 10 | 28 | 9 | 27 | 10 | 26 | 10 | 28 | 11 | 27
  Increase | 7331.62 (6411.996) | 5283.78 (4744.807) | 5731.61 (5064.881) | 4934.00 (4812.350) | 6793.00 (6076.280) | 5961.02 (5470.426) | 7572.53 (9023.363) | 6342.74 (5917.203) | 5863.90 (5274.304) | 7369.19 (6552.358) | 8389.80 (6625.523) | 6358.61 (5253.083)
  No Change: number analyzed (Participants) | 8 | 2 | 7 | 2 | 7 | 2 | 8 | 2 | 7 | 2 | 7 | 2
  No Change | 5283.54 (4043.599) | 5743.41 (2819.277) | 4216.93 (2660.723) | 6930.38 (5483.666) | 6412.49 (4323.454) | 5649.83 (1833.540) | 6158.33 (5186.584) | 6108.42 (1258.428) | 8118.69 (5998.806) | 4683.26 (7.859) | 4352.99 (3873.342) | 8688.22 (3272.243)
  <50% Reduction: number analyzed (Participants) | 56 | 24 | 55 | 24 | 53 | 21 | 55 | 21 | 50 | 22 | 56 | 23
  <50% Reduction | 6422.25 (6830.753) | 5449.38 (5289.323) | 6495.06 (5936.803) | 5356.63 (5359.524) | 6848.24 (6467.601) | 5315.31 (6041.242) | 7836.17 (8644.447) | 5399.55 (4159.097) | 8304.71 (8562.548) | 6567.55 (7807.345) | 7335.57 (7068.643) | 6481.35 (6132.009)
  50% to < 100% Reduction: number analyzed (Participants) | 6 | 0 | 8 | 0 | 7 | 0 | 8 | 0 | 6 | 0 | 5 | 0
  50% to < 100% Reduction | 2925.07 (3765.497) |  | 5352.66 (8413.472) |  | 5151.19 (6608.284) |  | 4892.41 (7615.700) |  | 7230.42 (9546.409) |  | 9795.94 (12602.08) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 5647.56 (1738.940) |  | 5510.19 (123.439) |  | 2265.42 (2731.172) |  | 731.08 |  | 533.76 (461.885) |  | 440.59 (225.383) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 2389.46 (964.418) |  | 2693.13 (1334.197) |  | 2482.52 (208.398) |  | 2450.90 (1729.041) |  | 2144.28 (1851.862) |  | 2896.76 (1518.588) |
  Overall | 6072.78 (6251.565) | 5374.40 (4875.645) | 5991.56 (5741.490) | 5195.78 (4999.201) | 6431.69 (6100.377) | 5677.37 (5562.787) | 7151.83 (8160.286) | 5928.95 (5068.858) | 7525.25 (7893.011) | 6926.73 (6941.824) | 7098.86 (7113.465) | 6502.50 (5540.461)

29. Secondary Outcome: Descriptive Statistics for Cigarettes Smoked Per Day (CPD) (Recall Data) in Day 1 and 8 (Respectively) by Study Group and Cigarette Consumption Categories
Description: Descriptive statistics for Cigarettes Smoked per Day (CPD) in Day 1 (Visit 2) and Day 8 (Visit 3) in Test and Control groups using recall data are presented. Subjects were sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing').
Time Frame: Day 1 (Visit 2) and Day 8 (Visit 3)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: cigarettes per day
Groups:
- Test (Visit 2): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Visit 2 (Day 1)
- Control (Visit 2): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Visit 2 (Day 1)
- Test (Visit 3): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Visit 3 (Day 8)
- Control (Visit 3): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Visit 3 (Day 8)
Arm/Group | Test (Visit 2) | Control (Visit 2) | Test (Visit 3) | Control (Visit 3)
Number analyzed (Participants) | 74 | 50 | 79 | 50
cigarettes per day
  Increase: number analyzed (Participants) | 10 | 27 | 10 | 28
  Increase | 15.6 (4.12) | 19.7 (8.52) | 16.1 (4.68) | 19.9 (8.47)
  No Change: number analyzed (Participants) | 6 | 2 | 8 | 2
  No Change | 19.5 (8.80) | 20.0 (0.00) | 17.6 (8.28) | 20.0 (0.00)
  <50% Reduction: number analyzed (Participants) | 48 | 21 | 52 | 20
  <50% Reduction | 18.4 (5.97) | 19.8 (6.96) | 18.2 (4.94) | 20.2 (6.36)
  50% to < 100% Reduction: number analyzed (Participants) | 6 | 0 | 6 | 0
  50% to < 100% Reduction | 16.0 (6.54) |  | 16.8 (5.85) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0
  100% Reduction | 12.5 (3.54) |  | 11.0 (2.83) |
  Missing: number analyzed (Participants) | 2 | 0 | 1 | 0
  Missing | 15.0 (7.07) |  | 20.0 |
  Overall | 17.7 (6.04) | 19.8 (7.64) | 17.6 (5.36) | 20.0 (7.43)

30. Secondary Outcome: Summary Statistics of Cigarettes Smoked Per Day (IVRS Data) by Study Group and Cigarette Consumption Categories on Days 1 Through 8
Description: Summary Statistics of Cigarettes Smoked per Day collected by IVRS Data method on Days 1 to 8 for Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
Time Frame: Daily during Baseline Period (Day 1 to Day 8)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: cigarettes per day
Groups:
- Test (Day 1): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Day 1
- Control (Day 1): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Day 1
- Test (Day 2): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Day 2
- Control (Day 2): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Day 2
- Test (Day 3): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Day 3
- Control (Day 3): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Day 3
- Test (Day 4): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Day 4
- Control (Day 4): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Day 4
- Test (Day 5): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Day 5
- Control (Day 5): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Day 5
- Test (Day 6): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Day 6
- Control (Day 6): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Day 6
- Test (Day 7): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Day 7
- Control (Day 7): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Day 7
- Test (Day 8): Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) Day 8
- Control (Day 8): Control Group (subjects continued ad libitum use of their own brand of tobacco products) Day 8
Arm/Group | Test (Day 1) | Control (Day 1) | Test (Day 2) | Control (Day 2) | Test (Day 3) | Control (Day 3) | Test (Day 4) | Control (Day 4) | Test (Day 5) | Control (Day 5) | Test (Day 6) | Control (Day 6) | Test (Day 7) | Control (Day 7) | Test (Day 8) | Control (Day 8)
Number analyzed (Participants) | 86 | 53 | 68 | 47 | 69 | 47 | 72 | 44 | 68 | 43 | 67 | 49 | 76 | 42 | 87 | 55
cigarettes per day
  Increase: number analyzed (Participants) | 11 | 29 | 9 | 25 | 7 | 24 | 9 | 26 | 9 | 23 | 8 | 25 | 10 | 19 | 11 | 29
  Increase | 16.5 (3.67) | 19.1 (8.04) | 15.4 (4.42) | 17.4 (8.39) | 17.0 (5.13) | 20.00 (8.66) | 17.0 (5.34) | 20.3 (8.49) | 15.8 (5.31) | 19.4 (9.63) | 15.8 (7.91) | 20.7 (9.82) | 15.4 (9.06) | 18.4 (8.75) | 17.5 (7.67) | 19.3 (8.58)
  No Change: number analyzed (Participants) | 8 | 2 | 7 | 2 | 8 | 2 | 8 | 1 | 7 | 1 | 8 | 2 | 8 | 2 | 8 | 2
  No Change | 17.4 (8.43) | 20.0 (0.00) | 18.7 (8.30) | 20.0 (0.00) | 17.4 (8.40) | 20.0 (0.00) | 17.6 (8.28) | 20.0 | 18.4 (8.52) | 20.0 | 17.1 (8.54) | 20.0 (0.00) | 17.5 (8.33) | 20.0 (0.00) | 17.3 (8.48) | 20.0 (0.00)
  <50% Reduction: number analyzed (Participants) | 56 | 22 | 43 | 20 | 43 | 21 | 44 | 17 | 43 | 19 | 43 | 22 | 47 | 21 | 56 | 24
  <50% Reduction | 19.1 (5.92) | 17.4 (7.12) | 17.9 (5.50) | 19.1 (6.48) | 17.3 (5.06) | 20.6 (6.45) | 18.8 (5.42) | 21.2 (7.06) | 17.8 (5.64) | 20.8 (8.30) | 17.9 (5.77) | 19.1 (5.77) | 18.9 (5.39) | 18.8 (6.74) | 18.6 (5.21) | 19.0 (6.87)
  50% to < 100% Reduction: number analyzed (Participants) | 7 | 0 | 5 | 0 | 7 | 0 | 8 | 0 | 7 | 0 | 4 | 0 | 7 | 0 | 8 | 0
  50% to < 100% Reduction | 18.4 (8.22) |  | 16.2 (5.85) |  | 19.1 (6.28) |  | 17.4 (5.66) |  | 18.6 (5.62) |  | 18.3 (8.88) |  | 17.4 (10.44) |  | 19.0 (5.86) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 8.5 (4.95) |  | 11.5 (4.95) |  | 8.5 (2.12) |  | 10.0 |  |  |  | 15.0 (0.00) |  | 11.5 (3.54) |  | 11.0 (5.66) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 15.0 (7.07) |  | 15.0 (7.07) |  | 15.5 (6.36) |  | 16.0 (5.66) |  | 17.0 (7.07) |  | 17.0 (7.07) |  | 21.0 (12.73) |  | 17.5 (10.61) |
  Overall | 18.2 (6.26) | 18.4 (7.49) | 17.3 (5.72) | 18.2 (7.41) | 17.2 (5.68) | 20.2 (7.46) | 18.1 (5.74) | 20.7 (7.79) | 17.6 (5.83) | 20.0 (8.87) | 17.4 (6.37) | 20.0 (7.96) | 18.0 (6.93) | 18.7 (7.48) | 18.2 (6.01) | 19.2 (7.63)

31. Secondary Outcome: Median Change From Baseline to End of Study for Urinary Total NNAL by Study Group
Description: Median change from baseline to End of Study for urinary total NNAL in Test and Control groups are presented. Baseline = Day 8 (Visit 3) values.
Time Frame: Day 8 (Visit 3) and End of Study (Day 36±1)
Population: Per-Protocol Population
Measure: Median (Inter-Quartile Range); unit: ng/g
Groups:
- Test (Change at End of Study/Early Term): Median change in Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) from Baseline to End of Study
- Control (Change at End of Study/Early Term): Median change in Control Group (subjects continued ad libitum use of their own brand of tobacco products) from Baseline to End of Study
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 87 | 55 | 87 | 55 | 87 | 55
ng/g | 472.893 [42.92 to 2072.61] | 395.108 [41.9 to 1524.88] | 444.709 [16.53 to 2851.85] | 476.795 [59.67 to 1558.82] | 5.448 [-564.08 to 1872.75] | 70.129 [-408.32 to 683.71]

32. Secondary Outcome: Median Change From Baseline to End of Study for Urinary Total NNAL by Study Group and Cigarette Consumption Categories
Description: Median Change from baseline to End of Study for urinary total NNAL in Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented. Baseline = Day 8 (Visit 3) values
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Median (Full Range); unit: ng/g
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 84 | 55 | 86 | 54 | 84 | 54
ng/g
  Increase: number analyzed (Participants) | 10 | 29 | 11 | 28 | 10 | 28
  Increase | 548.817 [103.304 to 1289.911] | 415.790 [75.406 to 1238.478] | 719.799 [252.923 to 1424.581] | 489.729 [59.671 to 1188.119] | 168.889 [-36.828 to 376.475] | 67.998 [-325.835 to 638.215]
  No Change: number analyzed (Participants) | 7 | 2 | 7 | 2 | 7 | 2
  No Change | 499.544 [132.328 to 843.698] | 789.559 [54.238 to 1524.880] | 376.087 [175.045 to 590.850] | 592.508 [68.451 to 1116.564] | 30.576 [-467.611 to 54.268] | -197.051 [-408.315 to 14.213]
  <50% Reduction: number analyzed (Participants) | 55 | 24 | 56 | 24 | 55 | 24
  <50% Reduction | 516.752 [42.916 to 2072.612] | 356.857 [41.901 to 1431.914] | 444.709 [18.574 to 2050.275] | 467.615 [84.686 to 1558.824] | 1.776 [-564.082 to 1208.177] | 73.507 [-111.025 to 683.712]
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 0
  50% to < 100% Reduction | 375.183 [57.698 to 979.102] |  | 263.677 [62.899 to 2851.852] |  | -48.425 [-365.303 to 1872.750] |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 158.649 [157.063 to 160.236] |  | 28.686 [16.528 to 40.844] |  | -129.963 [-140.535 to -119.392] |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 303.452 [124.886 to 482.019] |  | 268.140 [146.165 to 390.115] |  | -35.312 [-91.904 to 21.279] |
  Overall | 472.893 [42.916 to 2072.612] | 395.108 [41.901 to 1524.880] | 444.709 [16.528 to 2851.852] | 476.795 [59.671 to 1558.824] | 5.448 [-564.082 to 1872.750] | 70.129 [-408.315 to 683.712]

33. Secondary Outcome: Change From Baseline to End of Study Summary Statistics of Urinary Total NNAL (ng/g Creatinine) by Study Group and Cigarette Consumption Categories Over Visits
Description: Change from Baseline to End of Study summary statistics of urinary total NNAL (ng/g Creatinine) by Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented. Baseline = Visit 3 (Day 8) values.
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/g
Groups:
- Test (Change at End of Study/Early Term): Mean change in Test Group (subjects continued ad libitum use of their own brand of tobacco products and permitted ad libitum use of the test product [VBM-FG2 oral discs]) from Baseline to End of Study
- Control (Change at End of Study/Early Term): Mean change in Control Group (subjects continued ad libitum use of their own brand of tobacco products) from Baseline to End of Study
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 84 | 55 | 86 | 54 | 84 | 54
ng/g
  Increase: number analyzed (Participants) | 10 | 29 | 11 | 28 | 10 | 28
  Increase | 551.02 (318.270) | 440.36 (261.806) | 721.93 (327.377) | 538.09 (287.478) | 158.11 (140.443) | 92.60 (227.975)
  No Change: number analyzed (Participants) | 7 | 2 | 7 | 2 | 7 | 2
  No Change | 456.39 (275.603) | 789.56 (1039.900) | 389.46 (170.153) | 592.51 (741.128) | -66.92 (185.884) | -197.05 (298.772)
  <50% Reduction: number analyzed (Participants) | 55 | 24 | 56 | 24 | 55 | 24
  <50% Reduction | 535.46 (393.698) | 487.20 (378.047) | 614.61 (517.499) | 590.28 (451.453) | 88.22 (320.921) | 103.08 (170.772)
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 0
  50% to < 100% Reduction | 443.02 (343.687) |  | 592.73 (932.562) |  | 149.71 (713.457) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 158.65 (2.244) |  | 28.69 (17.194) |  | -129.96 (14.950) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 303.45 (252.531) |  | 268.14 (172.499) |  | -35.31 (80.032) |
  Overall | 507.43 (365.172) | 473.50 (347.581) | 586.29 (525.084) | 563.30 (376.309) | 81.33 (345.110) | 86.53 (209.749)

34. Secondary Outcome: Percent Change From Baseline to End of Study Summary Statistics of Urinary Total NNAL (%) by Study Group and Cigarette Consumption Categories Over Visits
Description: Percent change from Baseline to End of study summary statistics of urinary total NNAL (%) for Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
  Baseline = Visit 3 (Day 8) values.
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 84 | 55 | 86 | 54 | 84 | 54
percent change from baseline
  Increase: number analyzed (Participants) | 10 | 29 | 11 | 28 | 10 | 28
  Increase | 551.02 (318.270) | 440.36 (261.806) | 721.93 (327.377) | 538.09 (287.478) | 43.2 (49.11) | 31.7 (66.12)
  No Change: number analyzed (Participants) | 7 | 2 | 7 | 2 | 7 | 2
  No Change | 456.39 (275.603) | 789.56 (1039.900) | 389.46 (170.153) | 592.51 (741.128) | -0.3 (29.55) | -0.3 (37.46)
  <50% Reduction: number analyzed (Participants) | 55 | 24 | 56 | 24 | 55 | 24
  <50% Reduction | 535.46 (393.698) | 487.20 (378.047) | 614.61 (517.499) | 590.28 (451.453) | 17.6 (63.88) | 26.9 (48.80)
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 0
  50% to < 100% Reduction | 443.02 (343.687) |  | 592.73 (932.562) |  | 7.3 (80.69) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 158.65 (2.244) |  | 28.69 (17.194) |  | -82.0 (10.58) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 303.45 (252.531) |  | 268.14 (172.499) |  | -1.0 (25.53) |
  Overall | 507.43 (365.172) | 473.50 (347.581) | 586.29 (525.084) | 563.30 (376.309) | 15.4 (62.42) | 28.4 (57.66)

35. Secondary Outcome: Change From Baseline to End of Study Summary Statistics of Nicotine Equivalents (mg/g Creatinine) by Study Group and Cigarette Consumption Categories Over Visits
Description: Change from Baseline to End of Study summary statistics of urinary nicotine equivalents (mg/g creatinine) by Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
  Nicotine equivalents include nicotine and its 5 metabolites (cotinine, trans-3'-hydroxycotinine, trans-3'-hydroxycotinine-0-glucuronide, nicotine-N-glucuronide, and cotinine-N-glucuronide).
  Baseline = Visit 3 (Day 8) values.
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 80 | 50 | 79 | 48 | 74 | 46
mg/g
  Increase: number analyzed (Participants) | 10 | 27 | 11 | 24 | 10 | 23
  Increase | 18.24 (14.941) | 13.70 (7.870) | 24.84 (14.892) | 16.55 (6.791) | 6.77 (7.432) | 3.73 (5.932)
  No Change: number analyzed (Participants) | 6 | 1 | 6 | 2 | 6 | 1
  No Change | 8.75 (4.809) | 8.14 | 10.23 (3.053) | 13.62 (1.600) | 1.48 (3.418) | 6.61
  <50% Reduction: number analyzed (Participants) | 53 | 22 | 52 | 22 | 49 | 22
  <50% Reduction | 15.00 (9.726) | 14.77 (10.432) | 16.07 (11.551) | 18.07 (14.909) | 1.80 (9.214) | 3.29 (8.011)
  50% to < 100% Reduction: number analyzed (Participants) | 7 | 0 | 7 | 0 | 6 | 0
  50% to < 100% Reduction | 11.51 (6.995) |  | 16.62 (22.808) |  | 4.89 (20.082) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 1 | 0 | 1 | 0
  100% Reduction | 8.19 (1.870) |  | 7.41 |  | -2.11 |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 9.09 (1.956) |  | 8.81 (0.629) |  | -0.28 (2.585) |
  Overall | 14.32 (9.996) | 14.06 (8.973) | 16.60 (13.108) | 17.13 (11.092) | 2.59 (9.748) | 3.59 (6.886)

36. Secondary Outcome: Percent Change From Baseline to End of Study Summary Statistics of Nicotine Equivalents (%) by Study Group and Cigarette Consumption Categories Over Visits
Description: Percent change from Baseline to End of study summary statistics of urinary nicotine equivalents (%) for Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
  Nicotine equivalents include nicotine and its 5 metabolites (cotinine, trans-3'-hydroxycotinine, trans-3'-hydroxycotinine-0-glucuronide, nicotine-N-glucuronide, and cotinine-N-glucuronide).
  Baseline = Visit 3 (Day 8) values.
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 80 | 50 | 79 | 48 | 74 | 46
percent change from baseline
  Increase: number analyzed (Participants) | 10 | 27 | 11 | 24 | 10 | 23
  Increase | 18.24 (14.941) | 13.70 (7.870) | 24.84 (14.892) | 16.55 (6.791) | 62.5 (69.50) | 41.1 (72.40)
  No Change: number analyzed (Participants) | 6 | 1 | 6 | 2 | 6 | 1
  No Change | 8.75 (4.809) | 8.14 | 10.23 (3.053) | 13.62 (1.600) | 40.0 (55.51) | 81.1
  <50% Reduction: number analyzed (Participants) | 53 | 22 | 52 | 22 | 49 | 22
  <50% Reduction | 15.00 (9.726) | 14.77 (10.432) | 16.07 (11.551) | 18.07 (14.909) | 19.0 (61.98) | 27.6 (46.51)
  50% to < 100% Reduction: number analyzed (Participants) | 7 | 0 | 7 | 0 | 6 | 0
  50% to < 100% Reduction | 11.51 (6.995) |  | 16.62 (22.808) |  | 15.1 (93.59) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 1 | 0 | 1 | 0
  100% Reduction | 8.19 (1.870) |  | 7.41 |  | -22.1 |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 9.09 (1.956) |  | 8.81 (0.629) |  | -0.1 (28.42) |
  Overall | 14.32 (9.996) | 14.06 (8.973) | 16.60 (13.108) | 17.13 (11.092) | 25.2 (65.08) | 35.5 (60.54)

37. Secondary Outcome: Change From Baseline to End of Study Summary Statistics of S-PMA (ng/g Creatinine) by Study Group and Cigarette Consumption Categories Over Visits
Description: Change from Baseline to End of Study summary statistics of urinary S-phenyl mercapturic acid [S-PMA] (ng/g creatinine) by Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
  Baseline = Visit 3 (Day 8) values.
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 84 | 54 | 83 | 52 | 81 | 51
ng/g
  Increase: number analyzed (Participants) | 10 | 28 | 11 | 27 | 10 | 26
  Increase | 5731.61 (5064.881) | 4934.00 (4812.350) | 8389.80 (6625.523) | 6358.61 (5253.083) | 2410.02 (2986.346) | 1341.70 (2495.655)
  No Change: number analyzed (Participants) | 7 | 2 | 7 | 2 | 7 | 2
  No Change | 4216.93 (2660.723) | 6930.38 (5483.666) | 4352.99 (3873.342) | 8688.22 (3272.243) | 136.06 (3959.381) | 1757.84 (2211.423)
  <50% Reduction: number analyzed (Participants) | 55 | 24 | 56 | 23 | 55 | 23
  <50% Reduction | 6495.06 (5936.803) | 5356.63 (5359.524) | 7335.57 (7068.643) | 6481.35 (6132.009) | 875.52 (4755.856) | 903.68 (3218.825)
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 5 | 0 | 5 | 0
  50% to < 100% Reduction | 5352.66 (8413.472) |  | 9795.94 (12602.08) |  | 1941.73 (11042.40) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 5510.19 (123.439) |  | 440.59 (225.383) |  | -5069.60 (101.944) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 2693.13 (1334.197) |  | 2896.76 (1518.588) |  | 203.64 (184.391) |
  Overall | 5991.56 (5741.490) | 5195.78 (4999.201) | 7098.86 (7113.465) | 6502.50 (5540.461) | 903.49 (4985.072) | 1160.48 (2798.644)

38. Secondary Outcome: Percent Change From Baseline to End of Study Summary Statistics of S-PMA (%) by Study Group and Cigarette Consumption Categories Over Visits
Description: Percent change from Baseline to End of study summary statistics of urinary S-phenyl mercapturic acid [S-PMA] (%) for Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
  Baseline = Visit 3 (Day 8) values.
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 84 | 54 | 83 | 52 | 81 | 51
percent change from baseline
  Increase: number analyzed (Participants) | 10 | 28 | 11 | 27 | 10 | 26
  Increase | 5731.61 (5064.881) | 4934.00 (4812.350) | 8389.80 (6625.523) | 6358.61 (5253.083) | 50.0 (58.51) | 46.5 (76.26)
  No Change: number analyzed (Participants) | 7 | 2 | 7 | 2 | 7 | 2
  No Change | 4216.93 (2660.723) | 6930.38 (5483.666) | 4352.99 (3873.342) | 8688.22 (3272.243) | 16.1 (61.36) | 55.3 (75.66)
  <50% Reduction: number analyzed (Participants) | 55 | 24 | 56 | 23 | 55 | 23
  <50% Reduction | 6495.06 (5936.803) | 5356.63 (5359.524) | 7335.57 (7068.643) | 6481.35 (6132.009) | 19.9 (76.46) | 29.4 (66.18)
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 5 | 0 | 5 | 0
  50% to < 100% Reduction | 5352.66 (8413.472) |  | 9795.94 (12602.08) |  | 30.3 (123.78) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 5510.19 (123.439) |  | 440.59 (225.383) |  | -92.0 (3.91) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 2693.13 (1334.197) |  | 2896.76 (1518.588) |  | 6.7 (3.53) |
  Overall | 5991.56 (5741.490) | 5195.78 (4999.201) | 7098.86 (7113.465) | 6502.50 (5540.461) | 20.9 (76.27) | 39.1 (70.93)

39. Secondary Outcome: Change From Baseline to End of Study Summary Statistics of Carboxyhemoglobin (%) by Study Group and Cigarette Consumption Categories Over Visits
Description: Change from Baseline to End of Study summary statistics of blood carboxyhemoglobin (%) by Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented. Baseline = Visit 3 (Day 8) values.
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percent saturation of carboxyhemoglobin
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 87 | 55 | 87 | 55 | 87 | 55
percent saturation of carboxyhemoglobin
  Increase: number analyzed (Participants) | 11 | 29 | 11 | 29 | 11 | 29
  Increase | 6.62 (2.151) | 5.31 (1.627) | 5.97 (1.803) | 5.39 (1.786) | -0.65 (1.099) | 0.09 (1.178)
  No Change: number analyzed (Participants) | 8 | 2 | 8 | 2 | 8 | 2
  No Change | 5.68 (2.153) | 3.65 (2.192) | 5.00 (1.278) | 4.60 (1.414) | -0.68 (1.342) | 0.95 (0.778)
  <50% Reduction: number analyzed (Participants) | 56 | 24 | 56 | 24 | 56 | 24
  <50% Reduction | 5.40 (1.918) | 4.99 (2.184) | 5.11 (2.066) | 4.57 (1.847) | -0.29 (1.323) | -0.42 (0.986)
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 0
  50% to < 100% Reduction | 5.36 (2.159) |  | 3.21 (1.870) |  | -2.15 (0.952) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 4.45 (0.354) |  | 1.45 (0.212) |  | -3.00 (0.141) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 4.25 (2.333) |  | 3.65 (0.919) |  | -0.60 (1.414) |
  Overall | 5.53 (1.986) | 5.11 (1.897) | 4.91 (2.071) | 5.00 (1.821) | -0.61 (1.387) | -0.10 (1.118)

40. Secondary Outcome: Percent Change From Baseline to End of Study Summary Statistics of Carboxyhemoglobin (%) by Study Group and Cigarette Consumption Categories Over Visits
Description: Percent change from Baseline to End of study summary statistics of blood carboxyhemoglobin (%) for Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
  Baseline = Visit 3 (Day 8) values.
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 87 | 55 | 87 | 55 | 87 | 55
percent change from baseline
  Increase: number analyzed (Participants) | 11 | 29 | 11 | 29 | 11 | 29
  Increase | 6.62 (2.151) | 5.31 (1.627) | 5.97 (1.803) | 5.39 (1.786) | -7.6 (17.41) | 3.6 (27.54)
  No Change: number analyzed (Participants) | 8 | 2 | 8 | 2 | 8 | 2
  No Change | 5.68 (2.153) | 3.65 (2.192) | 5.00 (1.278) | 4.60 (1.414) | -4.0 (29.21) | 39.6 (45.07)
  <50% Reduction: number analyzed (Participants) | 56 | 24 | 56 | 24 | 56 | 24
  <50% Reduction | 5.40 (1.918) | 4.99 (2.184) | 5.11 (2.066) | 4.57 (1.847) | -3.7 (25.91) | -6.1 (18.12)
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 0
  50% to < 100% Reduction | 5.36 (2.159) |  | 3.21 (1.870) |  | -42.5 (18.66) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 4.45 (0.354) |  | 1.45 (0.212) |  | -67.5 (2.19) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 4.25 (2.333) |  | 3.65 (0.919) |  | -5.9 (30.05) |
  Overall | 5.53 (1.986) | 5.11 (1.897) | 4.91 (2.071) | 5.00 (1.821) | -9.3 (27.89) | 0.7 (25.53)

41. Secondary Outcome: Change From Baseline to End of Study Summary Statistics of Exhaled Carbon Monoxide (Ppm) by Study Group and Cigarette Consumption Categories Over Visits
Description: Change from Baseline to End of Study summary statistics of exhaled carbon monoxide (ppm) by Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
  Baseline = Visit 3 (Day 8) values.
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 88 | 55 | 87 | 55 | 87 | 55
ppm
  Increase: number analyzed (Participants) | 11 | 29 | 11 | 29 | 11 | 29
  Increase | 29.64 (12.118) | 20.59 (9.109) | 25.91 (8.860) | 20.21 (9.537) | -3.73 (10.248) | -0.38 (7.894)
  No Change: number analyzed (Participants) | 8 | 2 | 8 | 2 | 8 | 2
  No Change | 22.50 (9.562) | 11.50 (10.607) | 21.50 (9.957) | 18.50 (2.121) | -1.00 (9.798) | 7.00 (8.485)
  <50% Reduction: number analyzed (Participants) | 57 | 24 | 56 | 24 | 56 | 24
  <50% Reduction | 21.32 (10.133) | 20.96 (11.126) | 21.13 (10.091) | 19.08 (8.707) | -0.46 (8.466) | -1.88 (5.102)
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 0
  50% to < 100% Reduction | 20.63 (9.855) |  | 9.88 (6.081) |  | -10.75 (8.172) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 17.00 (4.243) |  | 4.00 (2.828) |  | -13.00 (1.414) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 18.50 (16.263) |  | 13.00 (8.485) |  | -5.50 (7.778) |
  Overall | 22.24 (10.491) | 20.42 (10.046) | 20.15 (10.410) | 19.65 (8.939) | -2.28 (9.175) | -0.76 (6.899)

42. Secondary Outcome: Percent Change From Baseline to End of Study Summary Statistics of Exhaled Carbon Monoxide (%) by Study Group and Cigarette Consumption Categories Over Visits
Description: Percent change from Baseline to End of study summary statistics of exhaled carbon monoxide for Test and Control groups sub-categorized by cigarette consumption categories obtained from End of Study ('Increase', 'No Change', >50% Reduction', '50 to <100% Reduction', '100% Reduction' and 'Missing') are presented.
  Baseline = Visit 3 (Day 8) values.
Time Frame: Day 8 (Visit 3) and Day 36 (Visit 7/End of Study)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Test (Visit 3) | Control (Visit 3) | Test (End of Study) | Control (End of Study) | Test (Change at End of Study/Early Term) | Control (Change at End of Study/Early Term)
Number analyzed (Participants) | 88 | 55 | 87 | 55 | 87 | 55
percent change from baseline
  Increase: number analyzed (Participants) | 11 | 29 | 11 | 29 | 11 | 29
  Increase | 29.64 (12.118) | 20.59 (9.109) | 25.91 (8.860) | 20.21 (9.537) | -7.0 (32.63) | 6.8 (58.17)
  No Change: number analyzed (Participants) | 8 | 2 | 8 | 2 | 8 | 2
  No Change | 22.50 (9.562) | 11.50 (10.607) | 21.50 (9.957) | 18.50 (2.121) | 6.6 (45.21) | 165.1 (226.09)
  <50% Reduction: number analyzed (Participants) | 57 | 24 | 56 | 24 | 56 | 24
  <50% Reduction | 21.32 (10.133) | 20.96 (11.126) | 21.13 (10.091) | 19.08 (8.707) | 6.0 (47.63) | -1.4 (40.74)
  50% to < 100% Reduction: number analyzed (Participants) | 8 | 0 | 8 | 0 | 8 | 0
  50% to < 100% Reduction | 20.63 (9.855) |  | 9.88 (6.081) |  | -49.2 (27.25) |
  100% Reduction: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  100% Reduction | 17.00 (4.243) |  | 4.00 (2.828) |  | -77.9 (11.11) |
  Missing: number analyzed (Participants) | 2 | 0 | 2 | 0 | 2 | 0
  Missing | 18.50 (16.263) |  | 13.00 (8.485) |  | -18.3 (25.93) |
  Overall | 22.24 (10.491) | 20.42 (10.046) | 20.15 (10.410) | 19.65 (8.939) | -3.1 (47.00) | 9.0 (66.04)

43. Secondary Outcome: Characterization of Subgroups Based on Change From Baseline in Total NNAL
Description: Statistical analyses on the number of subjects in subgroups based on urinary total NNAL change from baseline to the last visit are presented.
  Baseline = Visit 3 values.
Time Frame: Day 36 (Visit 7/End of Study) relative to the start of the baseline period (Visit 2/Day 1)
Population: Per-protocol
Measure: Count of Participants; unit: Participants
Groups:
- Test (ad Libitum VBM-FG2): Subjects were allowed to continue smoking their own brand of cigarettes ad libitum and were provided the option to use the test product (VBM-FG2 oral discs) also under ad libitum conditions)
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
Number analyzed (Participants) | 84 | 54
Participants
  Increase | 46 | 36
  Reduction | 38 | 18
Statistical Analysis 1: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); Null hypothesis = Test and Control groups will have equivalent number of subjects in subgroups based on urinary total NNAL change from baseline to end of study; Alternate hypothesis = Test and Control groups will NOT have equivalent number of subjects in subgroups based on urinary total NNAL change from baseline to end of study; Test type: Equivalence — Null hypothesis = Test and Control groups will have equivalent number of subjects in subgroups based on urinary total NNAL change from baseline to end of study; Alternate hypothesis = Test and Control groups will NOT have equivalent number of subjects in subgroups based on urinary total NNAL change from baseline to end of study; p = 0.1661, Cochran-Mantel-Haenszel; Probability = 0.1661 — Estimated value is the probability of observed distribution assuming the null hypothesis
Statistical Analysis 2: Comparison: Test (ad Libitum VBM-FG2) vs Control (no VBM-FG2); [analysis description as in outcome 43, analysis 1]; Test type: Equivalence — [test comment as in outcome 43, analysis 1]; p = 0.2139, Fisher Exact; Probability = 0.2139 — Estimated value is the probability of observed distribution assuming the null hypothesis

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the Informed Consent Form (ICF) by each subject until the end of the safety follow-up period, for a total of up to 9 weeks from Screening to End of Study per subject.
Description: One-hundred and fifty-seven (157) subjects were included in the Safety Population which included all subjects who tried the test product at least once during the study, including those subjects who participated only in the screening phase. Subjects were queried at each visit for any additional adverse events (AEs) or modifications to existing events.
Arm/Group | Test (ad Libitum VBM-FG2) | Control (no VBM-FG2)
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/62
Other Adverse Events (participants affected / at risk) | 25/92 | 7/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (ad Libitum VBM-FG2) (N=92) | Control (no VBM-FG2) (N=62)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Urogenital trichomoniasis (Infections and infestations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: COV-VER-01-13 Protocol Version 1 (2013-08-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT04079933/Prot_000.pdf
  • Study Protocol: COV-VER-01-13 Protocol Version 2 (2013-08-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT04079933/Prot_001.pdf
  • Statistical Analysis Plan (2013-10-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT04079933/SAP_002.pdf